CLINICAL TRIAL: NCT06393543
Title: International Registration of Isolated STIC: to Report and Investigate the Risk of Serous Peritoneal Carcinomatosis
Acronym: STICRISC
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17277
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: BRCA Mutation; Serous Tubal Intraepithelial Carcinoma; Ovarian Carcinoma; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Women with isolated STIC diagnosed between 2015 and the start of the study.
  Interventions: Other: No intervention, only registration
- Prospective cohort: Women with a newly diagnosed isolated STIC
  Interventions: Other: No intervention, only registration

INTERVENTIONS:
Other: No intervention, only registration — No intervention, only registration

SUMMARY:
To prospectively assess the incidence of peritoneal carcinomatosis for women with isolated STIC (serous tubal intraepithelial carcinoma). Moreover, to identify histopathological characteristics of STIC which are reproducible and associated to the risk of peritoneal carcinomatosis and to report the findings of additional diagnostics.

DETAILED DESCRIPTION:
Women with a BRCA pathogenic variant (PV) undergo a risk-reducing salpingo-oophorectomy (RRSO) to reduce their ovarian cancer risk of 17-44%. A residual risk for peritoneal cancer (PC) persists, with most patients having extensive tumour spread throughout the abdomen. Despite surgery and chemotherapy, the five-year survival rate of PC is only 14-30%. Recently it became apparent that PC is frequently preceded by a preinvasive serous tubal intraepithelial cancer (STIC) at RRSO. The entity STIC is often found conjointly with ovarian cancer, but can also be present as an isolated condition, mostly in high risk women. If this STIC is found at RRSO, the risk for PC was found to be 27.5% (95% CI, 15.6-43.9) after ten years whilst this risk was <1% without STIC. The pathophysiological mechanism of this association is not yet known and it is unknown which women with STIC are most at risk. Moreover, the additional value of diagnostics and management is unknown as data is lacking.

Objective: To prospectively assess the PC incidence for women with isolated STIC, to identify histopathological characteristics of STIC which are reproducible and associated to the risk of PC, and to report the findings of additional diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Bilateral salpingectomy (with or without oophorectomy)
* A serous tubal intraepithelial carcinoma at histopathological review

Exclusion Criteria:

* Invasive cancer at initial surgery or pathological examination (either macroscopic and/or microscopic)

Ages: 18 Years to 100 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: For the retrospective cohort: All women with STIC diagnosed between 2015 and start of the prospective study are identified. Data up until that time-point will be collected. At the end of the data collection follow-up will be updated on the women in the retrospective cohort.
  For the prospective cohort: All consecutive women with isolated STIC from participating centres are informed on the study and requested to participate.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2034-06 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
The risk for peritoneal carcinomatosis in women with isolated STIC | 10 years

SECONDARY OUTCOMES:
Risk factors | 5-10 years
  Risk for PC in relation to patient characteristics such as age at diagnosis and presence of a genetic pathogenic variant.
Histopathological characteristics | 5-10 years
  Identification of histopathological characteristics of STIC which are reproducible and associated to the risk of PC.
Additional diagnostics | 3 months
  To report findings at additional diagnostics (ie. imaging, staging surgery, CA125).

IPD SHARING:
Plan to Share IPD: Yes
In collaboration with participating centers upon reasonable request.